CLINICAL TRIAL: NCT04998058
Title: Autogenous Mesenchymal Stem Cell Culture-Derived Signalling Molecules as Enhancers of Bone Formation in Bone Grafting
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other); KU Leuven (Other); Rio Grande do Sul Brain Institute (InsCer) (Unknown)
Responsible Party: Principal Investigator, Eduardo Rolim Teixeira, DDS, Ph. D., Prof. Dr., Pontificia Universidade Católica do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Bone Graft-Exosomes Project
Record Dates: First submitted 2021-07-23; First posted 2021-08-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Bone Loss, Osteoclastic; Bone Loss, Alveolar; Alveolar Bone Loss; Alveolar Bone Atrophy; Grafting Bone
Keywords: bone; bone formation; bone graft; tissue engineering; stem cell; exosome; cell-free therapy
MeSH Terms: conditions — Bone Resorption; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled clinical trial, intra-individual (split-mouth design).
Who Masked: Participant, Outcomes Assessor
Masking Description: Bone tissue samples and image data allocation identified only by sequential numbers, not by name, for the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (conventional graft procedure), bone substitute and saline solution. (Placebo Comparator): one randomly assigned maxillary sinus grafted internally defined as control (bone substitute + saline solution) per subject.
  Interventions: Procedure: Maxillary sinus floor elevation grafting with synthetic bone substitute.
- Test (modified graft), bone substitute and concentrated culture medium (CM) (Experimental): one randomly assigned maxillary sinus grafted internally defined as test (bone substitute + concentrated culture medium) per subject.
  Interventions: Procedure: Maxillary sinus floor elevation grafting with synthetic bone substitute.

INTERVENTIONS:
Procedure: Maxillary sinus floor elevation grafting with synthetic bone substitute. — Bone augmentation at the floor of the maxillary sinus with bone substitutes.
  Other Names: Maxillary sinus lift bone grafting

SUMMARY:
This study aims to evaluate bone formation in grafts in terms of its quality (density), quantity (volume) and maturation obtained with the application of a tissue-engineered bone grafting compound containing concentrated autogenous cell-culture medium (CM) and a synthetic bone substitute. The present study was designed as an experimental prospective split-mouth randomized controlled clinical trial. After protocol approval by the Research Ethics Committee, a total of 20 consecutive participants in need of maxillary reconstruction aiming implant-supported oral rehabilitation will be invited to join the study. To collect autogenous adipose tissue-derived mesenchymal stem cells (hASCs), an outpatient lipoplasty procedure at the abdominal area of each patient will be performed. To isolate and expand hASCs from the lipoaspirate, specific cell culture protocols will be followed, resulting in cultured viable cells and their conditioned medium (CM). Cells and CM will be then separated by a sequence of filters and centrifugation, and isolated CM will be frozen. ELISA will analyze the presence of chemokines and their concentration in CM before grafting. Following pre-op surgical planning, both maxillary sinuses of each patient will be grafted internally applying a lateral window to each sinus. The bony floor of the test maxillary sinus will be augmented with synthetic bone substitute (BoneCeramic™ 1-2 mm) mixed with 10 to 15 ml of CM (test). The control site will receive bone substitute with saline. Lateral windows in both sinuses will be then closed with a collagen membrane (Bio-Gide™). After 6 months, first-stage implant surgery will be performed placing 6 implants in each patient. Registration of implant stability by manual torque wrench will be performed. Also, bone biopsies from each drilled implant site will be collected for histology, histomorphometry and immunohistochemistry (RT-PCR). Tomographic evaluation of the bone formation will include cone beam computed tomographies (CBCTs) at pre-operative [Baseline], 90 [T1] and 180 [T2 = implant placement] days for bone 3D image analysis.

DETAILED DESCRIPTION:
1. Aims and Hypothesis

   Based in previously reported studies and following a translational approach, a hypothesis that the paracrine effect linked to cultured autogenous growth factors and cytokines at physiologic concentrations acting locally in grafted sites might promote a faster and/or more efficient cell response and consequently induce a more significant/faster bone formation was considered. The presence of these molecules added to synthetic bone substitutes might act positively in terms of local cell recruitment (chemotaxis), proliferation, differentiation and bone protein synthesis. Also, recurrent biological hazards involved in conventional tissue-engineered cellular graft compounds, usually linked to the ex vivo manipulation of cells in terms of tumorigenicity, immunogenicity and the previously reported cell dedifferentiation phenomenon would be mitigated by the exclusion of the cell element of this process, as they are considered by some reports to present unpredictable mitotic behavior once artificially cultured. The present study aims to further extend this translational investigation following preclinical studies by the principal investigator, proposing a prospective randomized controlled clinical trial on the possible benefits associated with the application of a tissue-engineered bone graft compound containing concentrated autogenous cell-cultured medium (CM) and an hydroxylapatite/beta-tricalcium phosphate-based synthetic bone substitute (HP/β-TCP ceramic). Specific aims include analyses on the density of the newly formed calcified tissue by computed tomography (CBCTs), expression of specific immunohistochemical bone formation markers (RT-PCR) and histomorphometric bone quantity evaluation. In a split-mouth study model, the resultant bone formation after HP/β-TCP grafting with and without CM will be analyzed, compared and quantified at different time points.
2. Materials and Methods

2.1- Study design

A prospective split-mouth randomized controlled clinical trial was chosen as study design for the present investigation. After protocol approval by the Research Ethics Committee and registration at the clinical trials.gov platform, following CONSORT guidelines, 20 consecutive patients who seek maxillary oral rehabilitation at the Department of Prosthetic Dentistry of the School of Health and Life Sciences - PUCRS, Brazil, will be invited to participate in the present investigation.

2.2 - Lipoplasty and human adipose stem cells (hASCs) harvesting/culture.

For hASCs harvesting, an abdominal lipoplasty procedure will be proposed and performed following a signed informed consent. Under intravenous sedation and supplementary oxygen release with an oral catheter, along with local anesthesia, a standard surgical lipoplasty technique will be performed. As previously described, from this liposuction material, 25 to 30 ml of fat will be transferred into a 50 ml Falcon tube. The fat will be then washed by centrifugation (430Å~g 10 min), being the upper fat layer transferred into a new Falcon tube, where an equal volume of collagenase solution will be added to the mixture and incubated at 37°C in a water bath. After centrifugation, the upper fat layer will be discarded and the supernatant removed. The remaining cell pellet containing the hASCs will be resuspended with 15 ml of culture medium. After adding 15 ml of warm culture medium, the cell suspension will be transferred into a T175 culture flask. The hASCs will be incubated in a humidified environment at 37°C and 5% CO2. Then, the cell pellet will be resuspended in warm culture medium and seeded into new cell culture flasks.

2.3 - Concentrated culture medium (CM) preparation and analysis

Stem cell culture and CM preparation will be performed at a GMP certified facility for regenerative medicine products. At first, the surface antigen profiles of isolated hASCs at third passage will be characterized by flow cytometry. The presence of CD73, CD90, CD105 and CD44 markers and the absence of CD34, CD45, CD11b, CD19 and HLA-DR will be assessed to confirm the desired cell phenotype as recommended by protocols of the International Society of Cellular Therapy.[ Then, a sample of these cells will be also characterized by staining (Alizarin Red S) in accordance to the manufacturer's instructions. Cell expansion and CM will be generated following standard stem cell culture protocols. Before clinical use, CM will be examined not only for contamination with bacteria, fungi, or mycoplasmas but also for infection with viruses including hepatitis B and C, human immunodeficiency and human T-cell leukemia viruses. Then, CM will be properly cool-stored and sent to clinical application (up to 6 hours), to avoid long-term denaturation/inactivation of present signalling molecules, as previously suggested.

2.4 - Maxillary sinus floor elevation procedure

Under IV sedation and supplementary oxygen release with an oral catheter, along with local anesthesia, the maxillary bone will be grafted internally by drilling an access in the lateral maxillary sinus wall. Sinus membrane dissection with careful release and elevation will be also performed. Preoperative randomizing by computer-generated random numbers will be used to determine test and control sinuses for each patient. The bony floor of the maxillary sinus on the test site will be augmented with 4 to 5g of a synthetic bone substitute (BoneCeramic™ 1-2 mm) mixed with 10 to 15 ml of CM. The control site will receive similar amount of bone substitute embedded in 10 to 15 ml of saline solution. Patients will be released from hospital facility 2h after surgery. They will be instructed in postoperative hygiene and eating behavior. All patients will receive postoperative antibiotic and anti-inflammatory therapies.

2.5 - Implant placement and bone biopsies harvesting

After 6 months of healing, implant placement will follow routine surgical protocols as recommended by the implant manufacturer. Under local anesthesia, a mid-crestal linear incision and full-thickness flap will be performed with releasing incisions whenever necessary. Then, with a 16:1 contra-angle attached to a surgical unit and a trephine bur (Ø 3mm), the grafted area correspondent to the 2nd premolar, 1st and 2nd molar regions will be biopsied at both right and left sides of the maxilla (n=06 sites per patient), guided by a previously made acrylic resin surgical stent. Bone biopsies will be then divided in two segments, where one will be stored in 4% formaldehyde solution for histologic analysis and the other in Eppendorf vials with RNALater for RT-PCR analysis. Then, the sequence of implant surgical burs as recommended by the manufacturer will be followed for the placement of 6 to 8 implants per patient. Registration of primary stability at insertion will be done by both manual torque wrench and classified into three groups. A healing abutment will be then placed, and wound closure will be conducted with non-resorbable suture material A 6-month one-stage healing protocol will be adopted for all implants.

2.6 - CBCT image analysis

High-resolution CBCT images will be obtained at three different time-points as part of the treatment protocol, meaning at pre-operative bone graft [baseline], 90 [T1] and 180 [T2] days (implant placement pre-operative), aiming both pre-op surgical planning and post-op evaluation of the bone formation. The morphometric bone parameters will be calculated in 3D analysis according to the recommendations of the American Society for Bone and Mineral Research (ASBMR) as previously proposed, and statistical analysis will be used to identify the best parameter combinations aiming to differentiate trabecular bone into three bone categories: (i) sparse-related to a loose bone structure, (ii) intermediate-related to a well-structured trabecular bone, and (iii) dense bone types-related to a massive bone area with little space between the trabeculae.

2.7 - Histologic and histomorphometric analyses

Following removal of graft biopsies at implant placement, bone blocks containing the control and test bone sites will be shaped and decalcified with 5% HNO3. The blocks will dehydrate in a graded alcohol series, clarify with xylene and be embedded in resin. Then, the resin will be polymerised in a UV light chamber for 10h. Using a diamond micro saw, a total of three 3-μm-thick slices from each block will be ground transversely to each specimen long axis at 50, 100, and 150μm from their external portion. After this, routine staining with hematoxylin-eosin (HE), Azur II and Pararosaniline will be done aiming to differentiate between HP/β-TCP particles and newly formed bone. Microscopic analysis will be performed at 24X magnification using an optical stereo microscope connected to a digital camera. Image analysis will be performed using the ImageJ® software.

2.8 - Real-time polymerase chain reaction (RT-PCR)

Following the preparation of the collected graft biopsies for RNA extraction, real-time reverse transcriptase-polymerase chain reaction (RT-PCR) analysis will be applied to quantify alkaline phosphatase, vascular endothelial growth factor, Osteonectin, Osteopontin and type 1 collagen.

ELIGIBILITY:
Inclusion Criteria:

* patients >35 years-old.
* presenting highly atrophic fully edentulous maxilla (residual bone height <5 mm).
* In need of bilateral sinus floor augmentation aiming full mouth implant-supported rehabilitation.
* having teeth extraction at least 8 weeks prior to bone augmentation.

Exclusion Criteria:

* smokers, illicit drug users and alcohol daily consumers.
* patients with metabolic and/or systemic diseases leading to impaired healing (e.g. decompensated diabetes, leukocyte or coagulation disorders, immunosuppression).
* history of radiotherapy in the head or neck region.
* bisphosphonate-based therapy recipients.
* intolerant to general/local anesthesia.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in bone density and quantity | 0 (baseline), 90 and 180 days
  Comparative analysis (test vs. control) of the changes in bone density and quantity by cone beam computed tomography (CBCT).
Assessment of bone quantity | 180 days
  Histomorphometry analysis expressed in percentage of newly formed bone

SECONDARY OUTCOMES:
Presence of bone formation markers | 180 days
  RT-PCR assessing specific bone formation markers

OTHER OUTCOMES:
Assessment of bone substitute resorption rate | 180 days
  Resorption rate of bone substitute particles (test vs.control) compared by histologic analysis and histomorphometric analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo R Teixeira, DDS, Ph.D., Principal Investigator — Pontificia Universidade Católica do Rio Grande do Sul; Denise C Machado, MSc., Ph.D., Study Chair — Pontificia Universidade Católica do Rio Grande do Sul; Rogerio B Oliveira, DDS, Ph.D., Study Chair — Pontificia Universidade Católica do Rio Grande do Sul; Rosemary A Shinkai, DDS, Ph.D., Study Chair — Pontificia Universidade Católica do Rio Grande do Sul; Patricia Sesterheim, MSc, Ph.D., Study Chair — Institute of Cardiology of Rio Grande do Sul; Reinhilde Jacobs, DDS, Ph.D., Study Chair — KU Leuven
Locations (1):
- Pontificia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results will be informed in a publication.

REFERENCES:
- [Background] Cabreira CL, Fulginiti RL, Sesterheim P, Shinkai RSA, Teixeira ER. Effect of hyaluronic acid on paracrine signaling of osteoblasts from mesenchymal stromal cells: potential impact on bone regeneration. Clin Oral Investig. 2021 Jul;25(7):4571-4578. doi: 10.1007/s00784-020-03771-x. Epub 2021 Jan 7. PMID 33410999
- [Background] Teixeira ER, Boeckel D, Fulginiti R L, Shinkai R S A, Machado D. Mesenchymal stem cells and hyaluronic acid for bone grafting. Clinical Oral Implants Research, 2018, (29), 55-55.
- [Background] Boeckel DG, Sesterheim P, Peres TR, Augustin AH, Wartchow KM, Machado DC, Fritscher GG, Teixeira ER. Adipogenic Mesenchymal Stem Cells and Hyaluronic Acid as a Cellular Compound for Bone Tissue Engineering. J Craniofac Surg. 2019 May/Jun;30(3):777-783. doi: 10.1097/SCS.0000000000005392. PMID 30865107